CLINICAL TRIAL: NCT03161340
Title: Effect of Rapamycin on Pregnancy Rate of Patient With Recurrent Implantation Failure With Immunological Causes
Brief Title: Immunomodulatory Effects of Rapamycin on Pregnancy Rate of Patient With Recurrent Implantation Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mehdi Yousefi (Other)
Responsible Party: Sponsor-Investigator, Mehdi Yousefi, Tabriz University of Medical Sciences, Tabriz University of Medical Sciences
Organization: Tabriz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TabrizUMS-infertility-001
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Implantation Failure
Keywords: Recurrent Implantation Failure; Rapamycin; Pregnancy Rate
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Rapamycin group
  Interventions: Drug: Rapamycin
- Control group (No Intervention): Patients who do not receive any treatment despite a history of Recurrent Implantation Failure problem

INTERVENTIONS:
Drug: Rapamycin — Patients will take Rapamycin 2 days before IVF until 15 days after IVF
  Other Names: Treatment group
  Arms: Treatment group

SUMMARY:
Repeated implantation failure (RIF) is determined as failure to achieve pregnancy following at least 3 embryo transfers of high quality embryos in IVF cycles. Successful implantation and pregnancy depend on the activity of a variety of factors such as adhesion molecules, cytokines and immune cells.The process by which the foreign conceptus is accepted requires the appropriate function of regulatory T cells (Treg), which are known as the mediators of immune regulation. Tregs are capable of inducing maternal tolerance toward the fetus and their systemic expansion has been observed in early pregnancy. Furthermore, Th17 cells that play important roles in mounting inflammation are involved in the maintenance of pregnancy as a subset of effector T cells.The mammalian target of rapamycin (mTOR) inhibitors are immunosuppressive agents used after solid organ transplantation. Sirolimus as the most common mTOR inhibitor is able to effectively prevent allograft rejection and possesses significant antitumor properties. Pregnancy is a state of immunosuppression and the dysregulated immune responses has been observed in women with RIF. Accordingly, modulation of the immune system by an immunosuppressant drug may present an approach to overcome implantation failure. In this context, the use of Sirolimus might offer promise to achieve a better pregnancy outcome among women with implantation failure who undergo IVF. Based on previous findings, we hypothesized that Sirolimus may be beneficial for the improvement of pregnancy rate in women with IVF failure.

In the current study, we performe randomized phase II clinical trial to determine whether Sirolimus could be used as a bona fide treatment to increase the success rate of IVF in women with RIF of immune etiologies.A total 121 patients with a history of at least 3 RIF after IVF/ET cycles that will refer to Eastern Azerbaijan ACECR ART center, Alzahra Hospital of Tabriz University of Medical Sciences and Infertility Treatment center ACER Qom from July 2017 to June 2018 were select and enroll in this multicenter, randomized, double-blind, phase II study.

Normal ranges for Th17/Treg cell ratios establish using 50 normal fertile women who had a history of normal delivery by natural conception.

In patients with elevated Th17/Treg ratios, half of them treat with Sirolimus (Rapamune®; Pfizer, UK) and rest of patients not treat (control group). The patients in the treatment group will began Sirolimus 2 days prior to embryo transfer (ET) and will continue until the day of pregnancy test (15 day after ET), for a total of 17 days Sirolimus administe in a daily dose of 2mg.

ELIGIBILITY:
Inclusion Criteria:

* The patients selected for this study will be with elevated Th17/Treg ratio
* Enrolled patients will experience at least 3 times we have consecutive defeats implantation.
* Patients in the study will record their medical history do not have any type of immunotherapy.

Exclusion Criteria:

* Our criteria for exclusion of patients from the study include the following:
* Patients aged 20 years and above 41 years
* Patients or their spouse has abnormal karyotype or chromosomal and genetically disorders.
* Patients who have bleeding problems.
* Patients who have chronic disorders those are forced to use the specific drug.
* Patients who test HIV, hepatitis C virus (HCV) or hepatitis C virus (HBV) are positive.
* Patients who have a history of asthma and allergies to certain drugs.
* Patients who have abnormalities of the uterus

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Changes in Treg cells | 2 days before IVF until 15 days after IVF
  Flowcytometry
Changes in mRNA expression of cytokines related to Treg cells | 2 days before IVF until 15 days after IVF
  quantitative polymerase chain reaction (qPCR)
Changes in mRNA expression of cytokines related to Th17 cells | 2 days before IVF until 15 days after IVF
  quantitative polymerase chain reaction (qPCR)
Changes in secretion levels of cytokines related to Treg cells | 2 days before IVF until 15 days after IVF
  Elisa
Changes in secretion levels of cytokines related to Th17 cells | 2 days before IVF until 15 days after IVF
  Elisa
Changes in mRNA expression levels of transcription factors related to Th17 cells | 2 days before IVF until 15 days after IVF
  quantitative polymerase chain reaction (qPCR)
Changes in mRNA expression levels of transcription factors related to Treg cells | 2 days before IVF until 15 days after IVF
  quantitative polymerase chain reaction (qPCR)
Changes in expression levels of miRNAs | 2 days before IVF until 15 days after IVF
  quantitative polymerase chain reaction (qPCR)

SECONDARY OUTCOMES:
Pragnancy rate | 2 days before IVF until 15 days after IVF
  Beta-human Chorionic Gonadotrophin (ΒHCG) protein assay
Pregnancy Rate | 2 days before IVF until 15 days after IVF
  Ultrasonography
Live birth | After about 9 months of positive βhCG test
  The birth of a living child

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nouri, Ph.D, Study Director — SCARM institute; Mehdi Yousefi, Ph.D, Study Director — SCARM institute
Locations (2):
- Iran (2):
  - Qom ACECR ART Center, Qom
  - Estern Azarbaijan ACECR ART center, Tabriz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santos MA, Kuijk EW, Macklon NS. The impact of ovarian stimulation for IVF on the developing embryo. Reproduction. 2010 Jan;139(1):23-34. doi: 10.1530/REP-09-0187. PMID 19710204
- [Result] Sugiura-Ogasawara M, Suzuki S, Ozaki Y, Katano K, Suzumori N, Kitaori T. Frequency of recurrent spontaneous abortion and its influence on further marital relationship and illness: the Okazaki Cohort Study in Japan. J Obstet Gynaecol Res. 2013 Jan;39(1):126-31. doi: 10.1111/j.1447-0756.2012.01973.x. Epub 2012 Aug 13. PMID 22889462
- [Result] Calleja-Agius J, Muttukrishna S, Pizzey AR, Jauniaux E. Pro- and antiinflammatory cytokines in threatened miscarriages. Am J Obstet Gynecol. 2011 Jul;205(1):83.e8-16. doi: 10.1016/j.ajog.2011.02.051. Epub 2011 Feb 23. PMID 21514552
- [Result] Winger EE, Reed JL. Low circulating CD4(+) CD25(+) Foxp3(+) T regulatory cell levels predict miscarriage risk in newly pregnant women with a history of failure. Am J Reprod Immunol. 2011 Oct;66(4):320-8. doi: 10.1111/j.1600-0897.2011.00992.x. Epub 2011 Feb 14. PMID 21314851
- [Result] Ozkan ZS, Deveci D, Simsek M, Ilhan F, Risvanli A, Sapmaz E. What is the impact of SOCS3, IL-35 and IL17 in immune pathogenesis of recurrent pregnancy loss? J Matern Fetal Neonatal Med. 2015 Feb;28(3):324-8. doi: 10.3109/14767058.2014.916676. Epub 2014 May 22. PMID 24762139
- [Result] Winger EE, Reed JL, Ji X. First-trimester maternal cell microRNA is a superior pregnancy marker to immunological testing for predicting adverse pregnancy outcome. J Reprod Immunol. 2015 Aug;110:22-35. doi: 10.1016/j.jri.2015.03.005. Epub 2015 Apr 16. PMID 25965838
- [Result] Wang L, Harris TE, Roth RA, Lawrence JC Jr. PRAS40 regulates mTORC1 kinase activity by functioning as a direct inhibitor of substrate binding. J Biol Chem. 2007 Jul 6;282(27):20036-44. doi: 10.1074/jbc.M702376200. Epub 2007 May 17. PMID 17510057
- [Result] Nakagawa K, Kwak-Kim J, Ota K, Kuroda K, Hisano M, Sugiyama R, Yamaguchi K. Immunosuppression with tacrolimus improved reproductive outcome of women with repeated implantation failure and elevated peripheral blood TH1/TH2 cell ratios. Am J Reprod Immunol. 2015 Apr;73(4):353-61. doi: 10.1111/aji.12338. Epub 2014 Nov 14. PMID 25394810